CLINICAL TRIAL: NCT07199998
Title: Impact of the Use of Internal Menstrual Protections on Immunity and Vaginal Microbiota
Brief Title: Impact of Internal Menstrual Protections on Immunity and Vaginal Microbiota
Acronym: CUPS2
Status: Not yet recruiting | Type: Observational
Sponsor: Centre National de la Recherche Scientifique, France (Other)
Collaborators: Institut Alfred Fournier (Unknown)
Responsible Party: Principal Investigator, Samuel Alizon, Principal Investigator, Centre National de la Recherche Scientifique, France
Other Study IDs: 2024-A00597-40
Record Dates: First submitted 2025-08-20; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Sexual Transmitted Disease; Vaginosis, Bacterial; Mycosis; Urogenital Disease; HPV; Dysbiosis; Toxic Shock Syndrome; Menstrual Cup
Keywords: Menstrual cup; Dysbiosis; Menstrual health; Menstrual protection; Menstrual pad; Tampon; Immunity
MeSH Terms: conditions — Sexually Transmitted Diseases; Vaginosis, Bacterial; Mycoses; Urogenital Diseases; Dysbiosis; Shock, Septic | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal, cervical, urinary, and whole blood samples will be collected, each containing human and/or microbial DNA in varying proportions: vaginal and cervical samples provide both host and microbiota DNA, whole blood contains primarily human leukocyte DNA, while urine offers a mix of host epithelial and microbial DNA, though in lower quantity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tampon-only user: This group includes participants who have been using single-use tampons as their main form of menstrual protection in the past six months.
  Interventions: Other: Samples collection (whole blood, urine, vaginal and cervical cells)
- Cups-only user: This group includes participants who have used reusable menstrual cups as their main form of protection in the past six months.
  Interventions: Other: Samples collection (whole blood, urine, vaginal and cervical cells)
- External-only user: This group includes participants who have not used any internal menstrual products in the past six months, relying instead on external protection such as sanitary pads.
  Interventions: Other: Samples collection (whole blood, urine, vaginal and cervical cells)

INTERVENTIONS:
Other: Samples collection (whole blood, urine, vaginal and cervical cells) — During the clinical visit, samples will be collected from participants, including blood, urine, and vaginal and cervical cells. These samples will be used for a range of analyses, including determination of the vaginal microbiota composition and sequencing, cytokine profiling, and assessment of local immunity through flow cytometry using CyTOF technology. Urine samples will be analyzed for pollutants such as phthalates and bisphenol, while blood samples will be used for blood cell counts.

SUMMARY:
The availability, effectiveness, and safety of menstrual protection represent a key public health issue. However, research on women's menstrual and sexual health remains extremely limited. Whether societal or pathological, many hypotheses are emerging regarding the effects of menstrual protection products, yet little attention has been given to the products themselves, their societal role, or their physiological and pathological consequences. Internal menstrual products, such as tampons and menstrual cups, are widely used but are subject to limited regulatory oversight, and few studies have investigated their long-term effects on vaginal health.

This study aims to investigate how different types of menstrual protection influence vaginal microbiota, immune responses, and the recurrence of gynecological conditions such as bacterial vaginosis, mycosis, or dysbiosis. Biological samples (vaginal, cervical, urinary, and blood) will be collected to analyze vaginal microbiota composition and local immunity. Participants will be divided into three groups based on their main type of menstrual protection: menstrual cup users, tampon users, and external pad users. The study will compare these groups to assess potential differences in vaginal health and immune response related to menstrual product use.

DETAILED DESCRIPTION:
The aim of this study is to investigate potential links between the type of menstrual protection used and variations in vaginal health, including microbial composition, immune responses, and exposure to environmental pollutants.

The project consists of two complementary components:

- Epidemiological Study: An online survey will be conducted with 1,500 to 1,800 participants, collecting detailed information on the usage habits of menstrual protection products (such as menstrual cups, tampons, and external pads), as well as self-reported symptoms and history of urogenital infections. This dataset will allow for large-scale correlation analyses between menstrual hygiene practices and women's health indicators.

- Clinical Study:

A total of approximately 300 women will be recruited and divided into three groups based on their primary menstrual protection method:

Group 1: Menstrual cup users Group 2: Tampon users Group 3: External sanitary pad users

All clinical participants will undergo a gynecological examination and provide vaginal, cervical, urinary, and blood samples. These biological samples will be used for in-depth analysis across three main areas:

* Microbiology: studying the vaginal microbiota composition and identifying infectious or dysbiotic profiles.
* Immunology: assessing local immune responses, including cytokine levels and antibody titers.
* Toxicology: measuring exposure to potential environmental pollutants through menstrual product use.

Sequencing, immune profiling, pollutant quantification, and cytobacteriological screening will be conducted to evaluate potential differences between groups. These analyses aim to provide a better understanding of how menstrual protection methods may influence vaginal ecosystem balance, immune activity, and overall urogenital health.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study.
* Female, aged 18 to 49 years.
* In general good health, as determined by medical history.
* Covered by the national health insurance system.
* Willing to sign a written informed consent form.
* Has already experienced menstruation prior to the start of the study.
* No vaginal sexual intercourse within 72 hours before the study visit.
* Has had at least 6 menstrual periods in the past 12 months.

Exclusion Criteria:

* HIV infection.
* Positive diagnosis for chlamydia or syphilis at screening or within 4 weeks prior to screening.
* History of hormonal disorders or menstrual cycle irregularities.
* Metrorrhagia.
* Pregnancy or breastfeeding.
* Family members or close relatives of the clinical or scientific team.
* Treatment with any medication for chronic inflammatory disease or chronic conditions (e.g., cancer, arthritis, transplantation) within the past 12 months.
* Participation in an ongoing clinical trial.
* Receiving or having received antibiotic treatment within the 4 weeks prior to the study.
* Refusal to be informed in case of detected abnormalities.
* Indistinct use of both tampons and menstrual cups.
* Never having had vaginal penetrative intercourse.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population includes individuals of the female sex, aged 18 to 49 years, who have already experienced at least one menstrual period and meet the inclusion criteria. Participants are residents of the Île-de-France region and are recruited either through the Alfred Fournier Institute or via an online epidemiological survey.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Determine the effect of the use of internal menstrual products on the composition of the vaginal microbiota. | Samples will be stored at -80°C and metagenomics sequencing will be performed within 24 months after collection.
  To investigate potential differences in microbiota between study groups, the investigators will perform metagenomics next-generation sequencing on vaginal swabs.

SECONDARY OUTCOMES:
Comparison of the vaginal immune response of users and non-users of internal menstrual products | Samples for this purpose will be prepared for preservation immediately after collection. After preparation, they will be stored at -80°C and subsequently shipped for the analyses.
  Description of the cellular composition from vaginal and cervical samples (CyTOF technique) and measurement of vaginal cytokines.
  Since this is a cross-sectional study, all the measures are made at inclusion, i.e. at baseline.
Effect of the type of internal menstrual protections on the presence of pollutants in urine. | Urine samples will be stored at -80°C and analysed within 24 months after collection.
  Quantification of parabens and other pollutants in urine samples or other samples.

OTHER OUTCOMES:
Associations between the type of menstrual hygiene product used and sexually transmitted infections (STIs) | Statistical analyses will be performed after the last participant follow-up. They will be based on inclusion questionnaires. The time frame to evaluate the incidence of STIs will be the 12 months before inclusion.
  Retrospective epidemiological analyses will be performed using statistical modelling on the questionnaires filled in at the inclusion visit.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Alizon, Doctor in Biology, Principal Investigator — Centre National de la Recherche Scientifique, France
Locations (1):
- Institut Alfred Fournier, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided
Participants who wish to be informed about the results of the research will receive information in French about the scientific publications via a newsletter or posts on social media (e.g. mastodon).

REFERENCES:
- [Background] Tessandier N, Uysal IB, Elie B, Selinger C, Bernat C, Boue V, Grasset S, Groc S, Rahmoun M, Reyne B, Bender N, Bonneau M, Graf C, Tribout V, Foulongne V, Ravel J, Waterboer T, Hirtz C, Bravo IG, Reynes J, Segondy M, Murall CL, Boulle N, Kamiya T, Alizon S. Does exposure to different menstrual products affect the vaginal environment? Mol Ecol. 2023 May;32(10):2592-2601. doi: 10.1111/mec.16678. Epub 2022 Oct 4. PMID 36057782
- See also: French webpage of the study cohort — https://cups2.pages.in2p3.fr/cohorte/